CLINICAL TRIAL: NCT03544658
Title: Intervening Factors in Tooth Color Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Investigação em Bioquímica e Biologia Oral (Other)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BL 16000
Record Dates: First submitted 2018-04-30; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Tooth Color
Keywords: Tooth extrinsic stain; Tooth color; Dental prophylaxis; Visual shade guide; Dental spectrophotometer
MeSH Terms: interventions — Dental Prophylaxis

STUDY DESIGN:
Masking Description: Neither the patient, the investigator that made the color acquisition or the spectrophotometer had knowledge of tooth color assessed by the other person/method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental prophylaxis (Experimental): Visit 1: tooth color assessment (by patient, dentist and spectrophotometer) and professional dental prophylaxis Visit 2: tooth color assessment (by patient, dentist and spectrophotometer)
  Interventions: Procedure: Dental prophylaxis; Procedure: Tooth color assessment by the participant; Procedure: Tooth color assessment by the investigator; Procedure: Tooth color assessment with SpectroShade

INTERVENTIONS:
Procedure: Dental prophylaxis — Professional dental prophylaxis including dental scaling and dental polishing with prophylactic paste
Procedure: Tooth color assessment by the participant — Tooth color assessment using the VITA Classical shade guide. Assessment will be done with normal light conditions and with a light correcting device
Procedure: Tooth color assessment by the investigator — Tooth color assessment using the VITA Classical shade guide and the VITA Toothguide 3D Master. Assessment will be done with normal light conditions and with a light correcting device
Procedure: Tooth color assessment with SpectroShade — Tooth color assessment using SpectroShade (dental spectrophotometer). Color will be registered in VITA Classical and VITA Toothguide 3D Master and CIELab parameters

SUMMARY:
The aim of this study is to evaluate the influence of several factors (light, extrinsic stain removal and operator's experience) in tooth color assessment. Tooth color will be assessed by two different operators with visual shade guides under standardized light conditions and using a light correcting device (Smile Lite) or with a dental spectrophotometer in human subjects. Color measurement will be made before and 1 week after dental prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Capability to sign the informed consent
* Presence of upper teeth canines and central incisors, free of tooth decay, dental fillings, endodontic treatment or fixed rehabilitation
* Tooth color at least A3 in one of the included teeth
* Teeth should be possible to be subject to tooth color assessment with the predefined methods (color within the visual shade guides range)
* Absence of fixed orthodontic appliances or severe tooth structure anomalies

Exclusion Criteria:

* Pregnant patients
* Patients subjected to professional dental prophylaxis in less than 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Tooth color change determined before and after professional dental prophylaxis, assessed with visual shade guide (VITA Classical) | 1 week (measurements before and 1 week after dental prophylaxis)
  Tooth color will be determined prior to dental prophylaxis by the participant, investigator and spectrophotometer, using visual shade guide VITA Classical. 1 week after the intervention, the tooth color will be determined once again with the same protocol.
Tooth color change measured before and after professional dental prophylaxis, assessed with visual shade guide (VITA Toothguide 3D-Master) | 1 week (measurements before and 1 week after dental prophylaxis)
  Tooth color will be determined prior to dental prophylaxis by the investigator and dental spectrophotometer, using visual shade guide VITA Toothguide 3D-Master. 1 week after the intervention, the tooth color will be determined once again with the same protocol.
Tooth color change in CIELab system measured before and after professional dental prophylaxis | 1 week (measurements before and 1 week after dental prophylaxis)
  Tooth color in CIELab system will be determined by the conversion of VITA Classical shade guides in CIELab parameters assessed by the participant and investigator and by the spectroshade prior to professional dental prophylaxis. 1 week after the procedure tooth color will be determined once again with the same protocol.

SECONDARY OUTCOMES:
Agreement between operators in tooth color assessment with visual shade guides | Sequencial; repeated before and 1 week after intervention
  Comparison of tooth colors determined by the participant, investigator and spectrophotometer.
Influence of light conditions in tooth color assessment - change between determination with and without a light correcting device | Sequencial; repeated before and 1 week after intervention
  Tooth color determined by the participant and investigator with visual shade guides with two different light conditions: environmental light and assessment with a light correcting device (Smile Lite)

CONTACTS AND LOCATIONS:
Overall Officials: Duarte S Marques, PhD, DDS, Study Director — Grupo de Investigação em Bioquímica e Biologia Oral
Locations (1):
- Faculdade de Medicina Dentária, Universidade de Lisboa, Lisbon, Portugal